CLINICAL TRIAL: NCT06828380
Title: A Phase II Study of Immunotherapy With or Without Particle Beam Radiation Therapy in Patients With Advanced Hepatocellular Carcinoma Who Have Vascular Invasion: IOPT Study
Brief Title: A Study Comparing Immunotherapy Alone Versus Immunotherapy Combined With Radiotherapy in Patients With Hepatocellular Carcinoma (HCC) With Vascular Invasion
Acronym: IOPT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Bo Hyun Kim, Principal Investigator, National Cancer Center, Korea
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NCC2024-0308
Record Dates: First submitted 2025-01-27; First posted 2025-02-14 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): concurrent therapy of Immunotherapy based combination therapy and Proton beam radiation therapy
  Interventions: Radiation: Particle beam radiation therapy
- Arm B (No Intervention): concurrent therapy of Immunotherapy based combination therapy

INTERVENTIONS:
Radiation: Particle beam radiation therapy — The prescribed dose and fractionation for proton therapy to the PTV will be determined by the physician, taking into account the dose-volume constraints of normal tissues such as the liver and bowel.
  Arms: Arm A

SUMMARY:
In the present study, we aim to investigate the efficacy and safety of concurrent therapy of Immunotherapy based combination therapy and Radiotherapy in patients with advanced HCC showing macrovascular invasion.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Age >= 19 at the time of signing Informed consent form
3. Histological or clinical diagnosis of HCC based on the guidelines of the Korean Liver Cancer Association -National Cancer Center
4. Unresectable and/or locally advanced or metastatic disease showing major vascular invasion

   a. Presence of major vascular invasion on dynamic CT or dynamic MRI (1+2)
   * an intraluminal filling defect adjacent to the primary tumor in portal vein, hepatic vein, and/or inferior vena cava
   * an enhancement of the filling defect on arterial phase and a washout on portal/delayed phases
5. Having at least one measurable target lesion (per RECIST v1.1)

   a. Participants who received prior locoregional therapy (e.g., radiofrequency ablation, microwave ablation, transarterial chemoembolization, transarterial radioembolization, transarterial embolization, radiation therapy etc.) are eligible provided that other target lesion(s) have not been previously treated with locoregional therapy or the target lesion(s) within the field of locoregional therapy have subsequently progressed in accordance with RECIST v1.1.
6. Child-Pugh class A
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1
8. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 28 days prior to screening:

   1. Hemoglobin ≥ 8.0 g/dL
   2. Absolute neutrophil count (ANC) ≥ 1,000/mm3
   3. Platelet count ≥ 50,000/μL
   4. Total bilirubin < 3.0 mg/dL
   5. Serum albumin ≥ 2.8 g/dL
   6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 × the upper limit of normal (ULN)
   7. Prothrombin time in INR ≤ 1.8 × ULN
   8. Serum creatinine ≤ 2.0 × ULN or calculated creatinine clearance ≥ 40 mL/min (using the Cockcroft-Gault equation)
9. Documented virology status of hepatitis, as confirmed by screening tests for HBV and HCV

   a. Participants with HBV or HCV infection must be treated with antiviral therapy as per institutional practice.
10. Female participants of childbearing potential must agree to either remain abstinent or use effective contraception (with a failure rate of <1% per year) since signing of the informed consent form until at least 6 months after the last study drug administration.
11. Male participants must agree to remain abstinent or use a condom and refrain from donating sperm since signing of the informed consent form until at least 6 months after the last study drug administration.

Exclusion Criteria:

1. Fibrolamellar carcinoma or sarcomatoid carcinoma
2. Receipt of 2 or more prior systemic therapy for advanced HCC. Additional prior systemic therapies used as adjuvant or local therapy are allowed.
3. Receipt of other first-line systemic therapy than immune checkpoint inhibitor-based regimen
4. Receipt of prior radiation therapy to liver

   a. Participants are excluded if the potential radiation field overlaps with a previously irradiated area.
5. Receipt of locoregional therapy for HCC within 28 days prior to initiation of study treatment or non-recovery from complications due to the procedure (radiofrequency ablation, microwave ablation, cryoablation, trans-arterial embolization including chemo- and radio-embolization, or radiation therapy).

   a. A 7-day washout is permitted for palliative radiation to bone lesions
6. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, or multiple sclerosis with following exceptions:

   1. Patients with hypothyroidism stable on hormone replacement
   2. Controlled type 1 diabetes mellitus and on an insulin regimen
   3. Any chronic skin condition that does not require systemic therapy
7. Prior allogeneic stem cell or solid organ transplantation
8. Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to initiation of study treatment
9. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
10. Having active brain metastasis or leptomeningeal metastasis
11. Moderate to severe or intractable ascites
12. Presence of hepatic encephalopathy
13. History of malignancy other than HCC within 2 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate >90%)
14. Uncontrolled severe medical comorbidities, including significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to the initiation of study treatment, unstable arrhythmia, or unstable angina or any significant medical illness or abnormal laboratory findings that, in the investigator's judgement, would increase the risk to the participant associated with study participation
15. Female participants who are pregnant or breastfeeding or male or female participants of reproductive potential who are not willing to employ effective birth control from screening to 6 months after the last study drug administration
16. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2028-08-06 (Estimated); Study Completion 2028-08-06 (Estimated)

PRIMARY OUTCOMES:
PFS (Progression-free survival) | up to approximately 3 years
  PFS is defined as the time from the date of treatment initiation to the date of the first observation of progressive disease (PD) by the investigator according to RECIST v1.1 criteria or death from any cause.

SECONDARY OUTCOMES:
OS(overall survival) | up to approximately 3 years
  OS is defined as the time from the date of treatment initiation to the date of death from any cause.
TTP(Time to progression) | up to approximately 3 years
  TTP is defined as the time from the date of treatment initiation to the date of the first observation of PD by the investigator according to RECIST v1.1 criteria.
ORR(Objective response rate) | up to approximately 3 years
  ORR is defined as the proportion of participants whose best overall response is CR or PR as determined by the investigator according to RECIST v1.1 criteria.
DCR(Disease control rate) | up to approximately 3 years
  DCR is defined as the proportion of participants whose best overall response is a CR, PR, or SD as determined by the investigator according to RECIST v1.1 criteria.
DoR(Duration of response) | up to approximately 3 years
  DoR is defined as the time interval from the date of the first occurrence of a documented objective response (CR or PR, whichever occurs first) until the first date that disease progression or death is documented, whichever occurs first.
TTR(Time to response) | up to approximately 3 years
  TTR is defined as the time from the date of treatment initiation to the date of the first observation of a documented objective response (CR or PR, whichever occurs first).

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - National Cancer Center, Goyang
  - Samsung Medical Center, Seoul, Seoul

IPD SHARING:
Plan to Share IPD: Undecided